CLINICAL TRIAL: NCT03205969
Title: Pilot Study : Effects of Mobile Game for Chemotherapy Side Effect Education on Life Quality of Cancer Patients
Brief Title: Effects of Mobile Game on Life Quality of Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Principal Investigator, Jung Soon Jang, Professor,Division of Hemato-oncology, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: C2014147
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; chemotherapy side effect; mobile game
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Functional mobile game (Experimental): Functional mobile game for chemotherapy side effect education
  Interventions: Device: Functional mobile game

INTERVENTIONS:
Device: Functional mobile game — Functional mobile game for chemotherapy side effect education

SUMMARY:
The purpose of this study is to determine whether functional games can be used to improve the adherence and quality of life of breast cancer patients with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast cancer
* Receiving breast cancer chemotherapy
* Patients who are using a smartphone and agree to use a mobile functional game

Exclusion Criteria:

* Patient with intellectual disability
* Diagnosed with congenital genetic disease
* Patients with a history of acquired brain injury such as cerebral palsy
* Developmental disorders, including autism
* Patients with language or learning disabilities

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01-05 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Questionnaires (IPAQ) | overall assessment period (3 weeks)
  To obtain comparable estimates of physical activity

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | overall assessment period (3 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Jungsoon Jang, MD.PhD, Study Chair — Professor

REFERENCES:
- [Background] Touillaud M, Foucaut AM, Berthouze SE, Reynes E, Kempf-Lepine AS, Carretier J, Perol D, Guillemaut S, Chabaud S, Bourne-Branchu V, Perrier L, Tredan O, Fervers B, Bachmann P. Design of a randomised controlled trial of adapted physical activity during adjuvant treatment for localised breast cancer: the PASAPAS feasibility study. BMJ Open. 2013 Oct 28;3(10):e003855. doi: 10.1136/bmjopen-2013-003855. PMID 24165030
- [Background] Beutel ME, Weissflog G, Leuteritz K, Wiltink J, Haselbacher A, Ruckes C, Kuhnt S, Barthel Y, Imruck BH, Zwerenz R, Brahler E. Efficacy of short-term psychodynamic psychotherapy (STPP) with depressed breast cancer patients: results of a randomized controlled multicenter trial. Ann Oncol. 2014 Feb;25(2):378-84. doi: 10.1093/annonc/mdt526. Epub 2013 Dec 16. PMID 24347520
- [Background] Segrin C, Badger TA. Psychological and physical distress are interdependent in breast cancer survivors and their partners. Psychol Health Med. 2014;19(6):716-23. doi: 10.1080/13548506.2013.871304. Epub 2014 Jan 2. PMID 24383980
- [Background] DeNysschen CA, Burton H, Ademuyiwa F, Levine E, Tetewsky S, O'Connor T. Exercise intervention in breast cancer patients with aromatase inhibitor-associated arthralgia: a pilot study. Eur J Cancer Care (Engl). 2014 Jul;23(4):493-501. doi: 10.1111/ecc.12155. Epub 2013 Dec 2. PMID 24289215
- [Background] Carayol M, Romieu G, Bleuse JP, Senesse P, Gourgou-Bourgade S, Sari C, Jacot W, Sancho-Garnier H, Janiszewski C, Launay S, Cousson-Gelie F, Ninot G. Adapted physical activity and diet (APAD) during adjuvant breast cancer therapy: design and implementation of a prospective randomized controlled trial. Contemp Clin Trials. 2013 Nov;36(2):531-43. doi: 10.1016/j.cct.2013.09.016. Epub 2013 Oct 4. PMID 24096188
- [Background] Jung KW, Won YJ, Kong HJ, Oh CM, Seo HG, Lee JS. Cancer statistics in Korea: incidence, mortality, survival and prevalence in 2010. Cancer Res Treat. 2013 Mar;45(1):1-14. doi: 10.4143/crt.2013.45.1.1. Epub 2013 Mar 31. PMID 23613665
- [Background] Hwang SY, Chang SJ, Park BW. Does chemotherapy really affect the quality of life of women with breast cancer? J Breast Cancer. 2013 Jun;16(2):229-35. doi: 10.4048/jbc.2013.16.2.229. Epub 2013 Jun 28. PMID 23843858
- [Derived] Kim HJ, Kim SM, Shin H, Jang JS, Kim YI, Han DH. A Mobile Game for Patients With Breast Cancer for Chemotherapy Self-Management and Quality-of-Life Improvement: Randomized Controlled Trial. J Med Internet Res. 2018 Oct 29;20(10):e273. doi: 10.2196/jmir.9559. PMID 30578205